CLINICAL TRIAL: NCT00335270
Title: A Randomized, Prospective Study of the Efficacy, Safety and Tolerability of Two Doses of GW433908Ritonavir Given With Abacavir/Lamivudine Fixed Dose Combination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6692-05-12R1
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: HIV
Keywords: HIV Type 1
MeSH Terms: interventions — Ritonavir; abacavir; Lamivudine; abacavir, lamivudine drug combination

INTERVENTIONS:
Drug: fos-amprenavir calcium, ritonavir
Drug: abacavir/lamivudine as Epzicom

SUMMARY:
The purpose of this study is to evaluate the antiretroviral efficacy, safety, and tolerability of fos-amprenavir boosted with either of two doses of ritonavir (RTV) when administered in combination with ABC/3TC (abacavir/lamivudine, Epzicom®) FDC (fixed dose combination) in a once-daily regimen over 96 weeks in ART-naïve, HIV-infected adults

DETAILED DESCRIPTION:
The optimal long-term management of HIV-1 infection necessitates the chronic use of highly effective, well-tolerated antiretroviral (ARV) combination therapy, which ideally can preserve future treatment options. Current preferred standard treatment for HIV consists of a regimen composed of a protease inhibitor (PI) or a non-nucleoside reverse transcriptase inhibitor (NNRTI) plus 2 nucleoside reverse transcriptase inhibitors (NRTIs). A recent trend that may contribute to improving rates of treatment response is to use regimens with fewer pills and once daily dosing. This study is designed to assess two PI options that consist of four or five pills taken once daily - these options may also offer advantages in terms of metabolic consequences.

The primary objective of this multi-center, open-label, randomized, two-arm, pilot study is to evaluate the antiretroviral efficacy, safety, and tolerability (adverse events and metabolic profile) of fos-amprenavir (fAPV) boosted with either of two doses of ritonavir (RTV) when administered in combination with ABC/3TC (abacavir/lamivudine, Epzicom®) FDC (fixed dose combination) in a once-daily regimen over 48 weeks in ART-naïve, HIV-infected adults. Approximately 100 subjects will be enrolled from about 10 sites in the United States. Subjects must be >18 years of age, be ART-naïve (<7 days of prior therapy with any licensed or investigational ARV drugs) and have a plasma HIV-1 RNA>1,000 copies/mL. A CD4+ cell count >50 cells/mm3 was initially required for eligibility. Amendment 1 has dropped this as a requirement. Subjects will be stratified at entry according to their screening plasma HIV-1 RNA level (<100,000 copies/mL or >100,000 copies/mL). Eligible subjects will be randomized (1:1) to one of the following two treatment arms for 96 weeks; fAPV 1400 mg/RTV 100 mg QD plus ABC 600 mg/3TC 300 mg FDC QD (Treatment Arm A) or fAPV 1400 mg/RTV 200 mg QD plus ABC 600 mg/3TC 300 mg FDC QD (Treatment Arm B).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Male or Female 18 years of age or older
* Has plasma HIV-1 RNA (viral load) 1,000 or more copies/mL at screening
* Subject is antiretroviral-naïve ( less than 7 days of prior therapy with any agent
* Competency
* Not pregnant and willing to use effective birth control if applicable.

Exclusion Criteria:

* Inability to comply due to pre-existing mental, physical, or substance abuse disorder or other reason.
* Has active/acute CDC Clinical Category C event at screening.
* Has history of inflammatory bowel disease, gastrointestinal malignancy, intestinal ischemia, malabsorption or other gastrointestinal dysfunction.
* Females who are pregnant or breastfeeding.
* Has a serious medical condition, such as diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction, which in the opinion of the investigator would compromise the safety of the subject.
* Has ongoing clinically relevant pancreatitis or clinically relevant hepatitis at screening.
* Requires treatment with foscarnet, hydroxyurea or other agents with documented activity against HIV-1 in vitro within 28 days of study drug administration.
* Has an acute laboratory abnormality at screening that, in the opinion of the investigator, should preclude the subject's participation in the study. Any Grade 4 laboratory result would exclude a subject from study participation.
* Has required treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to screening, or has an anticipated need for such a treatment within the study period.
* Requires treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, vaccines, or interferons) within 28 days prior to screening or subject has received an HIV-1 immunotherapeutic vaccine within 90 days prior to screening.
* Has a history of allergy to any of the study drugs or any excipients therein.
* Is enrolled or plans to enroll in one or more investigational drug protocols, which may impact HIV RNA suppression.
* Requiring treatment with pharmacological agents for diabetes, or elevated triglycerides/cholesterol.
* Has an AST or ALT >5 times the upper limit of normal (ULN).
* Has an estimated creatinine clearance <50 mL/min via the Cockcroft-Gault method
* Subject requires treatment with any of the following medications within 28 days prior to study drug administration, or the anticipated need during the study: amiodarone, astemizole, bepridil, cisapride, dihydroergotamine, ergonovine, ergotamine, flecainide, halofantrine, lidocaine, lovastatin, methylergonovine, midazolam, pimozide, propafenone, quinidine, simvastatin, terfenadine, and triazolam, carbamazepine, dexamethasone, phenobarbital, phenytoin, primidone, rifampin, and St. John's Wort (hypericum perforatum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV 1 RNA <400 copies at week 48
Proportion of subjects who experience drug related discontinuations at Week 48

SECONDARY OUTCOMES:
Proportion of subjects who achieve plasma HIV 1 RNA<400 copies/mL at Weeks 24 and 96
Proportion of subjects who achieve plasma HIV-1 RNA <50 copies/mL at Weeks 24, 48, and 96.
Absolute values and change from baseline in plasma HIV-1 RNA and CD4+ cell counts at Weeks 24, 48, and 96.
Development and identification of genotypic resistance mutations and phenotypic resistance at virologic failure.
Incidence of Grades 2 to 4 AEs, treatment-limiting AEs, and serious adverse events (SAEs) over 24, 48, and 96 weeks.
Change from baseline in fat distribution as determined by percent change in body fat using whole body DEXA scans at Weeks 48, 72, and 96.
Change from baseline in subject's self-report of body fat distribution using the Body Image Questionnaire and the investigator's assessment of subject's body fat distribution using FRAM 2 PE (Grunfeld et al., 2003) at Weeks 48, 72, and 96.
Change from baseline in fasting lipids (total cholesterol, HDL cholesterol, direct LDL cholesterol, and triglycerides), fasting glucose and insulin measurements at Weeks 12, 24, 48, and 96.
Measurements of plasma APV trough concentrations at Weeks 4, 8, 24, and 48
To assess relationships between plasma APV trough concentrations and outcomes, including safety, efficacy and the development of resistance.
Adherence to each treatment regimen using pill counts of unused study drugs and subject self-assessment adherence questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hicks, MD, Principal Investigator — Duke University; Rafael E Campo, MD, Principal Investigator — University of Miami; Jason Flamm, MD, Principal Investigator — Medicine 4; Jeffrey Lennox, MD, Principal Investigator — Emory University; Rodger MacArthur, MD, Principal Investigator — Wayne State University; Jeffrey P Nadler, MD, Principal Investigator — Hillsborough County Health Department; John H. Schrank, MD, Principal Investigator — Greenville Hospital System; Louis Sloan, MD, Principal Investigator — North Texas Infectious Disease Consultants; Jeffrey Stephens, MD, Principal Investigator — Mercer University School of Medicine; David A Wohl, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

REFERENCES:
- [Background] Behrens G, Dejam A, Schmidt H, Balks HJ, Brabant G, Korner T, Stoll M, Schmidt RE. Impaired glucose tolerance, beta cell function and lipid metabolism in HIV patients under treatment with protease inhibitors. AIDS. 1999 Jul 9;13(10):F63-70. doi: 10.1097/00002030-199907090-00001. PMID 10416516
- [Background] Carpenter CC, Cooper DA, Fischl MA, Gatell JM, Gazzard BG, Hammer SM, Hirsch MS, Jacobsen DM, Katzenstein DA, Montaner JS, Richman DD, Saag MS, Schechter M, Schooley RT, Thompson MA, Vella S, Yeni PG, Volberding PA. Antiretroviral therapy in adults: updated recommendations of the International AIDS Society-USA Panel. JAMA. 2000 Jan 19;283(3):381-90. doi: 10.1001/jama.283.3.381. PMID 10647802
- [Background] Dube MP, Sprecher D, Henry WK, Aberg JA, Torriani FJ, Hodis HN, Schouten J, Levin J, Myers G, Zackin R, Nevin T, Currier JS; Adult AIDS Clinical Trial Group Cardiovascular Disease Focus Group. Preliminary guidelines for the evaluation and management of dyslipidemia in adults infected with human immunodeficiency virus and receiving antiretroviral therapy: Recommendations of the Adult AIDS Clinical Trial Group Cardiovascular Disease Focus Group. Clin Infect Dis. 2000 Nov;31(5):1216-24. doi: 10.1086/317429. Epub 2000 Nov 7. PMID 11073755
- [Background] Fung HB, Kirschenbaum HL, Hameed R. Amprenavir: a new human immunodeficiency virus type 1 protease inhibitor. Clin Ther. 2000 May;22(5):549-72. doi: 10.1016/S0149-2918(00)80044-2. PMID 10868554
- [Background] McComsey GA, Ward DJ, Hessenthaler SM, Sension MG, Shalit P, Lonergan JT, Fisher RL, Williams VC, Hernandez JE; Trial to Assess the Regression of Hyperlactatemia and to Evaluate the Regression of Established Lipodystrophy in HIV-1-Positive Subjects (TARHEEL; ESS40010) Study Team. Improvement in lipoatrophy associated with highly active antiretroviral therapy in human immunodeficiency virus-infected patients switched from stavudine to abacavir or zidovudine: the results of the TARHEEL study. Clin Infect Dis. 2004 Jan 15;38(2):263-70. doi: 10.1086/380790. Epub 2003 Dec 18. PMID 14699460
- [Background] Moore KH, Barrett JE, Shaw S, Pakes GE, Churchus R, Kapoor A, Lloyd J, Barry MG, Back D. The pharmacokinetics of lamivudine phosphorylation in peripheral blood mononuclear cells from patients infected with HIV-1. AIDS. 1999 Nov 12;13(16):2239-50. doi: 10.1097/00002030-199911120-00006. PMID 10563709
- [Background] Noble S, Goa KL. Amprenavir: a review of its clinical potential in patients with HIV infection. Drugs. 2000 Dec;60(6):1383-410. doi: 10.2165/00003495-200060060-00012. PMID 11152018
- [Background] Rodriguez-French A, Boghossian J, Gray GE, Nadler JP, Quinones AR, Sepulveda GE, Millard JM, Wannamaker PG. The NEAT study: a 48-week open-label study to compare the antiviral efficacy and safety of GW433908 versus nelfinavir in antiretroviral therapy-naive HIV-1-infected patients. J Acquir Immune Defic Syndr. 2004 Jan 1;35(1):22-32. doi: 10.1097/00126334-200401010-00003. PMID 14707788
- [Background] Tsiodras S, Mantzoros C, Hammer S, Samore M. Effects of protease inhibitors on hyperglycemia, hyperlipidemia, and lipodystrophy: a 5-year cohort study. Arch Intern Med. 2000 Jul 10;160(13):2050-6. doi: 10.1001/archinte.160.13.2050. PMID 10888979
- [Background] Walli R, Herfort O, Michl GM, Demant T, Jager H, Dieterle C, Bogner JR, Landgraf R, Goebel FD. Treatment with protease inhibitors associated with peripheral insulin resistance and impaired oral glucose tolerance in HIV-1-infected patients. AIDS. 1998 Oct 22;12(15):F167-73. doi: 10.1097/00002030-199815000-00001. PMID 9814858